CLINICAL TRIAL: NCT05333575
Title: The Effect of Lullaby and Classic Music to Prematures During Orogastric Tub Feeding on the Baby's Cerebral Oxygenization, Vital Findings and Comfort
Brief Title: Lullaby and Classic Music's Effect on Vital Findings and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sibel Küçükoğlu, Assoch Prof, Selcuk University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: SelcukUniversity
Record Dates: First submitted 2022-04-04; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Nutrition Disorder, Infant; Music; Preterm; Vital Signs
Keywords: preterm babies; cerebral oxygenation; lullabies; classical music
MeSH Terms: conditions — Infant Nutrition Disorders; Premature Birth

STUDY DESIGN:
Intervention Model Description: Research 28-34 preterm babies with gestational age hospitalized in the 2nd and 3rd level intensive care unit of Selcuk University Medical Faculty Hospital in Konya, Turkey. As a result of the power analysis, it was determined that the inclusion of 45 preterm infants in the study would provide sufficient sample size based on the two-sided hypothesis, 1.392 effect size, 0.05 margin of error and 0.95 power. Since the study period coincided with a period of uncertainties such as the Covid 19 pandemic, it was foreseen that there may be a loss in the number of babies included in the groups, and the sample number was increased by 10%, and the study was completed with a total of 51 premature babies (maternal voice group: 17, control group 17, classical music group 17).Babies of mothers who agreed to participate in the study were randomly assigned to the experimental and control groups. Simple randomization method was used in the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group: Lullaby (Experimental): The mothers in this group sang lullabies to their babies next to the incubator during feeding.
  Interventions: Behavioral: Lullaby
- Experimental Group: Classic Music (Experimental): Babies in this group were listened to classical music during feeding.
  Interventions: Behavioral: Classic music
- Control Group (No Intervention): Premature newborns in the control group were fed according to the routine of the clinic and no intervention was performed other than routine practice.

INTERVENTIONS:
Behavioral: Lullaby — The mothers in this group were asked to sing a lullaby while their babies were fed with an orogastric tube. Mothers were released on lullabies. They were encouraged to sing the lullaby they knew or loved the most. The mother was given a sound decibel meter. Mothers were asked to do an application before going to the baby. It was taught that the number of sound decibels should not exceed 40 decibels while singing a lullaby. Later, the mother was taken to the baby's incubator at feeding time. She was seated in a chair. The working status of the decibel meter was checked and given to the mother. When the feeding started, the mother started singing lullabies and continued to sing until the feeding was finished. Attention was paid to aseptic techniques during all procedures. A single mother was asked to sing a lullaby at each feeding, and the baby of the mother who sang only a lullaby was included in the study.
  Arms: Experimental Group: Lullaby
Behavioral: Classic music — The babies in this group were given classical music recitals during feeding. The classical music piece Mozart-Baby Smart was preferred because it was seen to be used in the literature (Keidar 2014). Mozart-Baby Smart was loaded into the music player by the researcher before the feeding process. Before feeding, the decibel meter was disinfected by surface disinfectant and placed on sterile sponge in an incubator 10 cm away from the baby's head. The music player was turned on, not exceeding 40 decibels, by adjusting the decibel meter at the time of starting the feeding, and classical music was continued during the feeding. When the feeding was finished, the music player was turned off and the incubator was taken out. Attention was paid to acetic techniques during all procedures. Ambient sounds were tried to be controlled as much as possible so that the baby would not be affected by different sounds when listening to classical music.
  Arms: Experimental Group: Classic Music

SUMMARY:
In the study, lullabies and classical music played to preterm babies during orogastric tube feeding; It will be tried to determine the effect on cerebral oxygenation level, vital signs and comfort levels.

DETAILED DESCRIPTION:
In the literature, there are many studies on prematurity pain and its relief. Although the vital signs and comfort levels of infants were examined in many applications for infants hospitalized in the neonatal intensive care unit, no study was found in which the cerebral oxygenation levels of infants were evaluated by NIRS by listening to lullabies and classical music to premature infants. There is no study in the literature examining cerebral oxygenation, vital signs and comfort parameters together during orogastric tube feeding, which is frequently used in preterm infants. For this reason, in this study, lullabies and classical music played to preterm babies during orogastric tube feeding; It will be tried to determine the effect on cerebral oxygenation level, vital signs and comfort levels. It is thought that the study will present new data to the literature and will lead many researches.

ELIGIBILITY:
Inclusion Criteria:

* Being at 28-34 weeks of gestation,
* Stability (in terms of cerebral oxygenation, pain and vital signs) during enrollment,
* Not having any additional diagnosis other than the diagnosis of prematurity,
* Indication of bolus feeding with an orogastric tube,

Exclusion Criteria:

* Congenital anomaly in the baby
* Diagnosed hearing impairment in the baby
* Having a history of an invasive procedure (such as a surgical operation) that will disrupt the baby's long-term comfort and cause pain
* The baby is receiving oxygen therapy or the baby is on mechanical ventilation
* Any history of disease affecting cerebral oxygenation (such as intraventricular hemorrhage, neonatal convulsions).

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Newborn Information Form | First measurement - Before intervention
  This form was developed by the researcher using the literature (Loewy et al 2013, Caparros-Gonzalez et al 2018, Azarmnejad et al 2015, Alipour et al 2013). The form was composed of questions including introductory information about the baby, gestational age, postnatal age, gender, birth weight (gr), weight on the day of the intervention, type of delivery, 1st and 5th min apgar score.
Regional brain oxygen saturation (rSO2) levels | First measurement - one minute before the baby is fed
  The form prepared by the researcher; It was prepared in such a way that physiological parameters such as baby's rSO2 levels were recorded. The form is designed to record twice, 1 minute before the baby is fed and immediately after the feeding is completed.
Heart rate (minute) | First measurement - one minute before the baby is fed
  The form prepared by the researcher; It was prepared in such a way that physiological parameters such as heart rate (min) were recorded. The form is designed to record twice, 1 minute before the baby is fed and immediately after the feeding is completed.
Oxygen saturation (%SpO2) | First measurement - one minute before the baby is fed
  The form prepared by the researcher; It was prepared in such a way that physiological parameters such as Oxygen saturation (%SpO2) were recorded.. The form is designed to record twice, 1 minute before the baby is fed and immediately after the feeding is completed.
Body temperature (°C) | First measurement - one minute before the baby is fed
  The form prepared by the researcher; It was prepared in such a way that physiological parameters such as baby's body temperature (°C) were recorded. The form is designed to record twice, 1 minute before the baby is fed and immediately after the feeding is completed.
Respiratory rate (min) | First measurement - one minute before the baby is fed
  The form prepared by the researcher; It was prepared in such a way that physiological parameters such as baby's respiratory rate (min) were recorded. The form is designed to record twice, 1 minute before the baby is fed and immediately after the feeding is completed.
COMFORTneo Scale | First measurement - one minute before the baby is fed
  The scale is a Likert type scale developed to determine the pain, distress, sedation and comfort needs of newborns followed in the intensive care unit. Ambuel et al. created the Comfort Scale in 1992 to evaluate the distress of children receiving mechanical ventilator support in pediatric intensive care units. Van Dijk et al. revised the scale in 2009 and made the validity and reliability of the COMFORTneo scale only to measure newborn behavior without vital parameters. The Turkish validity and reliability of the scale was performed by Kahraman et al. in 2014. The lowest score that can be obtained from the Newborn Comfort Behavior Scale is 6, and the highest score is 30. High scores indicate that the baby is not comfortable and needs interventions to provide comfort.

SECONDARY OUTCOMES:
Regional brain oxygen saturation (rSO2) levels | Second measurement - immediately after feeding
  The form prepared by the researcher; It was prepared in such a way that physiological parameters such as Oxygen saturation (%SpO2) were recorded.. The form is designed to record twice, 1 minute before the baby is fed and immediately after the feeding is completed.
Heart rate (minute) | Second measurement - immediately after feeding
  The form prepared by the researcher; It was prepared in such a way that physiological parameters such as heart rate (min) were recorded. The form is designed to record twice, 1 minute before the baby is fed and immediately after the feeding is completed.
Oxygen saturation (%SpO2) | Second measurement - immediately after feeding
  The form prepared by the researcher; It was prepared in such a way that physiological parameters such as Oxygen saturation (%SpO2) were recorded.. The form is designed to record twice, 1 minute before the baby is fed and immediately after the feeding is completed.
Body temperature (°C) | Second measurement - immediately after feeding
  The form prepared by the researcher; It was prepared in such a way that physiological parameters such as baby's body temperature (°C) were recorded. The form is designed to record twice, 1 minute before the baby is fed and immediately after the feeding is completed.
Respiratory rate (min) | Second measurement - immediately after feeding
  The form prepared by the researcher; It was prepared in such a way that physiological parameters such as baby's respiratory rate (min) were recorded. The form is designed to record twice, 1 minute before the baby is fed and immediately after the feeding is completed.
COMFORTneo Scale | Second measurement - immediately after feeding
  The scale is a Likert type scale developed to determine the pain, distress, sedation and comfort needs of newborns followed in the intensive care unit. Ambuel et al. created the Comfort Scale in 1992 to evaluate the distress of children receiving mechanical ventilator support in pediatric intensive care units. Van Dijk et al. revised the scale in 2009 and made the validity and reliability of the COMFORTneo scale only to measure newborn behavior without vital parameters. The Turkish validity and reliability of the scale was performed by Kahraman et al. in 2014. The lowest score that can be obtained from the Newborn Comfort Behavior Scale is 6, and the highest score is 30. High scores indicate that the baby is not comfortable and needs interventions to provide comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Kucukoglu, PhD, Study Chair — Selcuk University
Locations (2):
- Turkey (Türkiye) (2):
  - Selcuk University, Konya
  - Sibel Kucukoglu, Konya

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Background] Keidar HR, Mandel D, Mimouni FB, Lubetzky R. Bach music in preterm infants: no 'Mozart effect' on resting energy expenditure. J Perinatol. 2014 Feb;34(2):153-5. doi: 10.1038/jp.2013.138. Epub 2013 Nov 14. PMID 24232665
- [Background] Loewy J, Stewart K, Dassler AM, Telsey A, Homel P. The effects of music therapy on vital signs, feeding, and sleep in premature infants. Pediatrics. 2013 May;131(5):902-18. doi: 10.1542/peds.2012-1367. Epub 2013 Apr 15. PMID 23589814
- [Background] Caparros-Gonzalez RA, de la Torre-Luque A, Diaz-Piedra C, Vico FJ, Buela-Casal G. Listening to Relaxing Music Improves Physiological Responses in Premature Infants: A Randomized Controlled Trial. Adv Neonatal Care. 2018 Feb;18(1):58-69. doi: 10.1097/ANC.0000000000000448. PMID 29045255
- [Background] Azarmnejad E, Sarhangi F, Javadi M, Rejeh N. The Effect of Mother's Voice on Arterial Blood Sampling Induced Pain in Neonates Hospitalized in Neonate Intensive Care Unit. Glob J Health Sci. 2015 Apr 19;7(6):198-204. doi: 10.5539/gjhs.v7n6p198. PMID 26153174
- [Background] Alipour Z, Eskandari N, Ahmari Tehran H, Eshagh Hossaini SK, Sangi S. Effects of music on physiological and behavioral responses of premature infants: a randomized controlled trial. Complement Ther Clin Pract. 2013 Aug;19(3):128-32. doi: 10.1016/j.ctcp.2013.02.007. Epub 2013 May 9. PMID 23890458
- [Background] van Dijk M, Roofthooft DW, Anand KJ, Guldemond F, de Graaf J, Simons S, de Jager Y, van Goudoever JB, Tibboel D. Taking up the challenge of measuring prolonged pain in (premature) neonates: the COMFORTneo scale seems promising. Clin J Pain. 2009 Sep;25(7):607-16. doi: 10.1097/AJP.0b013e3181a5b52a. PMID 19692803
- [Background] Kahraman A, Başbakkal Z, Yalaz M, 2014. Yenidoğan Konfor Davranış Ölçeği'nin Türkçe geçerlik ve güvenirliği. Uluslararası Hakemli Hemşirelik Araştırmaları Dergisi, 1, 2, 1-11.
- [Derived] Bagli E, Kucukoglu S, Soylu H. The Effect of Lullabies and Classical Music on Preterm Neonates' Cerebral Oxygenation, Vital Signs, and Comfort During Orogastric Tube Feeding: A Randomized Controlled Trial. Biol Res Nurs. 2024 Apr;26(2):181-191. doi: 10.1177/10998004231202404. Epub 2023 Sep 22. PMID 37737114